CLINICAL TRIAL: NCT05604118
Title: Platelet Enzymatically Oxidized Phospholipids (eoxPL) Characterisation in a Healthy Cohort on and Off Aspirin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SMREC16/02
Record Dates: First submitted 2022-10-20; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Platelet Dysfunction Due to Aspirin
Keywords: platelets; phospholipids; aspirin
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin supplemented (Experimental)
  Interventions: Drug: Aspirin
- Off aspirin (No Intervention)

INTERVENTIONS:
Drug: Aspirin — 1 week of aspirin supplementation prior to sampling
  Arms: Aspirin supplemented

SUMMARY:
Healthy volunteers (n = 28) were recruited from the workplace (14 male, 14 female; age range 20-50 years). Ethical approval, which included informed consent, was from Cardiff University, Schools of Medicine and Dentistry Research Ethics Committee (SMREC16/02). Following a 2-week period free from non-steroidal anti-inflammatory drugs (NSAIDs), peripheral blood was obtained and platelets isolated. Participants were commenced on aspirin 75 mg once daily for seven days and then provided a repeat blood sample. Following a 2-month period, participants were invited to repeat samples pre- and post-aspirin, and again a third time 2 months later.

ELIGIBILITY:
Inclusion Criteria:

* two-week washout period from any non-steroidal anti-inflammatory drugs (NSAIDs) use.
* Ability to take aspirin 75 mg once daily for seven days and sampled thereafter, before stopping the aspirin.
* Willingness to repeat this process after two months and four months of the initial sampling date.

Exclusion Criteria:

* Recent NSAID use

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Platelet EoxPL differences in amounts (ng) as measured by liquid chromatography with tandem mass spectrometry | 4 months
  Samples on and off aspirin will be quantified for the 47 most common eoxPL species (as described by Slatter et al, Cell Metabolism 23, 930-944, May 10, 2016) using established liquid chromatography with tandem mass spectrometry (LC-MS/MS). Differences in amounts on and off aspirin will be quantified and tested for statistical significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Geraint Evans Cardiovascular Research Building, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No